CLINICAL TRIAL: NCT04894825
Title: A Phase I, Multi-center, Open-label, Single-dose Escalation and Expansion, Dose Escalation and Expansion Combination With Chemotherapy Study Evaluating the Safety, Tolerability and Pharmacokinetic Profile of M108 Monoclonal Antibody in Patients With Advanced Unresectable Solid Tumors in China
Brief Title: Safety, Tolerability and Pharmacokinetic Profile of M108 Monoclonal Antibody in Patients With Advanced Unresectable Solid Tumors in China
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: FutureGen Biopharmaceutical (Beijing) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M108-Ⅰ
Record Dates: First submitted 2021-05-12; First posted 2021-05-20 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Advanced Unresectable Solid Tumors
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Cohort (Experimental): Monotherapy: Five dose levels of M108 will be tested according to an accelerated titration method followed by a conventional 3 + 3 study design.
  Combined with chemotherapy: Three dose levels of M108 will be tested by a conventional 3 + 3 study design.
  The dose-limiting toxicity (DLT) will be assessed from the first administration to the end of the first cycle (21 days).
  Interventions: Drug: M108
- Dose Expansion Cohort (Experimental): Once the effective dose has been determined, 1~2 expansion cohorts will be opened to evaluate the efficacy and safety of the selected dose.
  Interventions: Drug: M108

INTERVENTIONS:
Drug: M108 — Monotherapy: Accelerated titration method, IV infusion Q3W; Conventional 3 + 3 study design, IV infusion Q3W. (21-day cycles) Combined with chemotherapy: Conventional 3 + 3 study design, IV infusion Q3W. (21-day cycles)
  Other Names: Chemotherapy
  Arms: Dose Escalation Cohort
Drug: M108 — IV infusion Q3W. (21-day cycles)
  Other Names: Chemotherapy.
  Arms: Dose Expansion Cohort

SUMMARY:
M108 is a monoclonal antibody specific for gastric and gastroesophageal adenocarcinomas. The aim of this phase I study is to establish safety and Tolerability of different Dosage regimen in patients With Advanced Unresectable Solid Tumors in China.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Advanced Unresectable solid tumors proven by histology
3. At least 1 measurable site of the disease according RECIST 1.1 criteria
4. ECOG performance status (PS) 0-1
5. Life expectancy > 3 months
6. Age ≥ 18 years and ≤75 years
7. Adequate haematological function; absolute neutrophil count ≥1.5 x 109/L; white blood cell count ≥3.0 x 109/L; platelets ≥100 x 109/L; haemoglobin ≥9 g/dL.
8. Adequate coagulation function; international normalized ratio ( INR) ≤ 1.5 x upper limit of normal (ULN), or activated partial thromboplastin time (APTT) ≤ 1.5 x ULN.
9. Adequate hepatic function; bilirubin ≤1.5 x ULN, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) ≤2.5 x ULN.
10. Adequate renal function; creatinine ≤1.5 x ULN, or reatinine clearance rate ≥60 mL/minute calculated.

Exclusion Criteria:

1. Previous received or planned to be vaccinated with 2019-nCoV vaccine or other vaccines within 3 months prior to the start of study treatment or during the study or within 3 months after the end of the study;
2. Previous radiotherapy within 4 weeks prior to the start of study treatment. (if palliative radiotherapy was given to bone metastatic side peripherally and the patient recovered from acute toxicity was allowed).
3. Previous anti-tumor therapy within 4 weeks prior to the start of study treatment.
4. Previous major operation within 8 weeks prior to the start of study treatment.
5. Prior severe allergic reaction or intolerance to a monoclonal antibody, including humanised or chimeric antibodies.
6. Symptomatic cerebral metastases.
7. Uncontrolled or severe illness.
8. Known human immunodeficiency virus infection or known symptomatic hepatitis
9. Other clinically significant disease which may have adversely affected the safe delivery of treatment within this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From enrollment until 28+7 days after the last dose
  defined by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE V5.0)
Maximum Tolerated Dose | 21 days
  MTD

SECONDARY OUTCOMES:
Maximum measured plasma concentration of M108 | From enrollment until 28 days after the last dose
  Cmax
Time to maximum plasma concentration of M108 | From enrollment until 28 days after the last dose
  Tmax
Half-life of M108 | From enrollment until 28 days after the last dose
  T1/2
Immunogenicity profile of M108 | From enrollment until 28 days after the last dose
  Blood samples will be collected from subjects post treatment for assessment to detect the presence of anti-drug antibodies(ADA).
Objective Response Rate | From first dose to disease progression , death or end of study，an average of 1 year
  ORR
Progression free survival | From first dose to disease progression , death or end of study，an average of 1 year
  PFS

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China